CLINICAL TRIAL: NCT00145210
Title: A Double-Blind, Randomized, Placebo- and Active-Controlled, Forced Titration Study Evaluating the Effects of Nebivolol on Blood Pressure and Heart Rate in African American Patients With Hypertension
Brief Title: Safety and Efficacy of Nebivolol in the Treatment of Hypertension in African Americans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Bertek Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB310
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension
Keywords: Nebivolol
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Atenolol

INTERVENTIONS:
Drug: Nebivolol and Atenolol

SUMMARY:
The purpose of this study is to evaluate the effects of nebivolol on blood pressure and heart rate in African American patients with hypertension.

DETAILED DESCRIPTION:
Despite the established benefits of beta-blockers, their use is limited by their side effect profile and by a perception of reduced efficacy in certain populations such as African Americans (Amudha, 2003). This is a double-blind, randomized, placebo and active-controlled, multi-center, parallel group, forced titration study. Patients will be stratified across all treatment arms by age, gender, and diabetes status (history of diabetes mellitus vs no history of diabetes mellitus). The study consists of 3 periods: screening run-in, double-blind, randomized, forced titration and double-blind, washout period (only for patients who complete the double-blind, forced titration period and who are not participating in the long-term follow-up study). After a 14-28 day, single-blind, placebo controlled, run-in period, which includes washout (if applicable), eligible patients will be randomized to one of 3 treatment regimens for approximately 12 weeks.

This study will test the safety and efficacy of Nebivolol in the treatment of African American patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* African Americans with stage 1-2 hypertension

Exclusion Criteria:

* Recent myocardial infarction or stroke
* Contraindications to beta-blocker therapy or stopping prior antihypertensive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Blood pressure
Heart Rate

SECONDARY OUTCOMES:
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Betty S. Riggs, MD, MBA, Study Director — Mylan Pharmaceuticals Inc
Locations (1):
- Mylan Pharmaceuticals Inc., Morgantown, West Virginia, United States